CLINICAL TRIAL: NCT00002839
Title: PHASE II STUDY ON LARYNX PRESERVATION COMPARING INDUCTION CHEMOTHERAPY AND RADIOTHERAPY VERSUS ALTERNATING CHEMO-RADIOTHERAPY IN RESECTABLE HYPOPHARYNX AND LARYNX CANCERS
Brief Title: Combination Chemotherapy Plus Radiation Therapy To Preserve the Larynx in Patients With Cancer of the Hypopharynx or Larynx
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-24954
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Head and Neck Cancer
Keywords: stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Fluorouracil; Neoadjuvant Therapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells and allow doctors to preserve the part of the body where the cancer started. It is not yet known which regimen of cisplatin and fluorouracil combined with radiation therapy is more effective in treating resectable cancer of the hypopharynx or larynx.

PURPOSE: Randomized phase III trial to compare the effectiveness of two regimens of cisplatin and fluorouracil combined with radiation therapy in preserving the larynx in patients who have resectable cancer of the hypopharynx or larynx.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare relapse-free survival and larynx preservation in patients with resectable hypopharyngeal or laryngeal cancer treated with sequential vs alternating cisplatin and fluorouracil and radiotherapy.
* Compare the health-related quality of life in patients treated with these regimens.
* Compare the cost-effectiveness of these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by performance status, disease site, tumor stage, node stage, and center.

Patients are randomized to one of two treatment arms. Both groups may receive either conventional radiotherapy in single daily fractions, 5 days per week, for 7 weeks (option 1) or hyperfractionated radiotherapy in 2 daily fractions, 5 days per week, for 4-5 weeks (option 2), according to institutional policy.

* Arm I: Patients receive cisplatin and fluorouracil every 3 weeks. Patients with a complete or partial response on day 42 receive 2 additional courses of chemotherapy followed by 7 weeks of radiotherapy beginning on day 80. After radiotherapy, patients with a complete remission enter follow-up; those with a partial remission proceed to surgery. Patients with stable or progressive disease proceed immediately to surgery with or without postoperative radiotherapy.
* Arm II: Patients receive cisplatin and fluorouracil every 3 weeks for 4 courses. Patients treated on radiotherapy option 1 are evaluated 2 months after completion of radiotherapy; those with a complete remission enter follow-up while all others proceed to surgery. Patients treated on option 2 are evaluated on day 42; those with a partial or complete response complete chemoradiotherapy and are then evaluated and treated like option 1 patients. Patients with stable or progressive disease on day 42 proceed to surgery with or without a third course of chemotherapy on week 7.

Patients are followed every 3 months for 3 years and at least every 6 months thereafter.

PROJECTED ACCRUAL: A total of 564 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven squamous cell carcinoma of the head and neck, including:

  * Stage III/IV cancer of the glottic or supraglottic larynx

    * Eligible T4 tumor defined as:

      * Bulging the valleculae
      * Bulging the hyothyroid membrane
      * Minimal thyroid cartilage invasion or suspicion of invasion on imaging
  * Stage II/III/IV cancer of the pyriform sinus or of the hypopharyngeal aspect of the aryepiglottic fold (with or without extension to postcricoid area)

    * No massive destruction of the thyroid cartilage
    * No continuity between primary tumor and a lymph node
* Operable on first attempt (as assessed by head and neck surgeon) by classical total laryngectomy with or without partial pharyngectomy

  * No requirement for extended surgery (circumferential pharyngolaryngectomy)
  * No tumor suitable for partial (functional) surgery or requiring extended surgery that necessitates any kind of flap for closure
  * No N2c tumor unless no requirement for bilateral resection of internal jugular veins
* Measurable or evaluable disease by panendoscopy and CT scan or MRI

  * Esophagoscopy required
  * Bronchofiberscopy recommended
* No requirement for tracheotomy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* WHO 0-2

Hematopoietic:

* WBC at least 4,000/mm^3

Hepatic:

* Bilirubin no greater than 2.0 times normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Other:

* No medical, psychological, or geographical condition that precludes study compliance
* No serious nonmalignant systemic disease
* No second malignancy except:

  * Carcinoma in situ of the cervix
  * Adequately treated nonmelanomatous skin cancer
* No poor nutritional status unlikely to be restored to fair status within 3 weeks
* No contraindication to CT scan or general anesthesia

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior anticancer biologic therapy

Chemotherapy

* No prior anticancer chemotherapy

Endocrine therapy

* No prior anticancer endocrine therapy

Radiotherapy

* No prior anticancer radiotherapy

Surgery

* See Disease Characteristics

Other

* No other prior anticancer therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 1996-07; Primary Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Lefebvre, MD, Study Chair — Centre Oscar Lambret; Jean-Claude Horiot, MD, PhD, Study Chair — Centre Georges Francois Leclerc
Locations (20):
- Belgium (2):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - Universitair Ziekenhuis Antwerpen, Edegem
- France (10):
  - CHR de Besancon - Hopital Jean Minjoz, Besançon
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier Universitaire de Dijon, Dijon
  - Centre de Lutte Contre le Cancer, Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Regional et Universitaire de Lille, Lille
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Centre Antoine Lacassagne, Nice
  - Hopital Charles Nicolle, Rouen
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
- Rambam Medical Center, Haifa, Israel
- Italy (3):
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Milano (Milan)
  - Ospedale Civile Monselice, Monselice, Padova
  - Azienda Ospedaliera "Santa Maria Degli Angeli", Pordenone
- Netherlands (3):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Leiden University Medical Center, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

REFERENCES:
- [Result] Lefebvre JL, Rolland F, Tesselaar M, Bardet E, Leemans CR, Geoffrois L, Hupperets P, Barzan L, de Raucourt D, Chevalier D, Licitra L, Lunghi F, Stupp R, Lacombe D, Bogaerts J, Horiot JC, Bernier J, Vermorken JB; EORTC Head and Neck Cancer Cooperative Group; EORTC Radiation Oncology Group. Phase 3 randomized trial on larynx preservation comparing sequential vs alternating chemotherapy and radiotherapy. J Natl Cancer Inst. 2009 Feb 4;101(3):142-52. doi: 10.1093/jnci/djn460. Epub 2009 Jan 27. PMID 19176454
- [Result] Lefebvre J, Horiot J, Rolland F, et al.: Phase III study on larynx preservation comparing induction chemotherapy and radiotherapy versus alternating chemoradiotherapy in resectable hypopharynx and larynx cancers. EORTC protocol 24954-22950. [Abstract] J Clin Oncol 25 (Suppl 18): A-LBA6016, 303s, 2007.
- [Derived] Bottomley A, Tridello G, Coens C, Rolland F, Tesselaar ME, Leemans CR, Hupperets P, Licitra L, Vermorken JB, Van Den Weyngaert D, Truc G, Barillot I, Lefebvre JL. An international phase 3 trial in head and neck cancer: quality of life and symptom results: EORTC 24954 on behalf of the EORTC Head and Neck and the EORTC Radiation Oncology Group. Cancer. 2014 Feb 1;120(3):390-8. doi: 10.1002/cncr.28392. Epub 2013 Oct 25. PMID 24452673